CLINICAL TRIAL: NCT00209404
Title: Iodixanol in Multidetector-Row Computed Tomography-Coronary Angiography (MDCT-CA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DXV407
Record Dates: First submitted 2005-08-18; First posted 2005-09-21 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Coronary Artery Disease
Keywords: MDCT; Coronary Artery; Heart Rate; Image Quality; Diagnostic Quality
MeSH Terms: conditions — Coronary Artery Disease | interventions — iodixanol

INTERVENTIONS:
Drug: Iodixanol 320 mg I/Ml

SUMMARY:
Image quality in coronary artery computed tomography is influenced by the heart rate variation during the examination. The purpose of this clinical trial is to investigate the change in heart rate following injection of a contrast medium called Visipaque™ (iodixanol). Image quality and diagnostic quality of the examination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with low to moderate suspicion of coronary artery disease referred for retrospective electrocardiogram (ECG)-gated multidetector row computed tomography coronary angiography and with a heart rate >75 beats per minute (bpm) will be included.

Exclusion Criteria:

* Subjects who take medications that slow down the heart rate or present cardiac arrhythmia at rest will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-07

PRIMARY OUTCOMES:
Change in mean heart rate

SECONDARY OUTCOMES:
Image quality
Diagnostic quality
Overall diagnostic information
Frequency and intensity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Antonini, Study Director — GE Healthcare
Locations (1):
- Amersham Health S.A., Vélizy-Villacoublay, France